CLINICAL TRIAL: NCT00023439
Title: Study of the Performance of Several Nucleic Acid Amplification Methodologies in the Diagnosis and Management of Active TB
Brief Title: TBTC NAA Study: Pilot Study of Surrogate Markers for Outcome of TB Treatment
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Stefan Goldberg, CDC
Other Study IDs: CDC-NCHSTP-2530; NAA TBTC
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-06

CONDITIONS: Tuberculosis
Keywords: tuberculosis; TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: Nucleic Acid Amplification Methods for diagnosis — no intervention

SUMMARY:
This is a pilot study to evaluate the performance of several nucleic acid amplification methodologies in the diagnosis and management of active tuberculosis

DETAILED DESCRIPTION:
This study evaluates potential surrogate markers of treatment failure and relapse as a substudy of ongoing Tuberculosis Trials Consortium (TBTC) disease treatment studies. After enrollment is complete, specimens from cases of treatment failure and relapse will be evaluated in comparison to control samples to measure the prognostic value of the following tests: 1) quantitative rRNA in 2-month sputum to predict relapse, 2) MTB 85B mRNA to detect reactivation, 3) 1- to 4-month NAA and broth culture tests to predict relapse, 4) mRNA, rRNA and DNA at and after end of therapy to predict relapse, 5)sputum rRNA and blood DNA to detect recurrence during prodrome, 6) sputum rRNA compared to cultures to diagnose "paradoxical reactions," 7) compare blood DNA to cultures at end of induction and end of treatment, 8) compare accuracies of different NAA assays and standard cultures, 9) determine MTD rRNA assay positive to negative conversion time, 10) characterize quality and quantity of sputum over time in relation to culture and clinical outcome, 11) assess ability of clinical, radiographic, and microbiologic risk factors to predict treatment failure and relapse.

ELIGIBILITY:
Inclusion Criteria:

1. (1) Enrollment in another TBTC treatment study, or (2) Suspected or culture-confirmed pulmonary TB (designated "NAA2"). Acceptable as indicators of suspected tuberculosis -- culture -- will be a positive AFB smear or a positive M. tuberculosis NAA test for MTB.
2. (For NAA2 cases only): Collection of a sputum specimen for NAA processing, obtained in the interval from 14 days before, to 17 days after the start of anti-tuberculosis treatment.
3. Physician recommendation and patient willingness to receive tuberculosis therapy as described in another TBTC treatment trial or in accordance with CDC/ATS recommendations as outlined below:

   Induction phase therapy will be initiated with 4-drugs (isoniazid, PZA, rifamycin and either ethambutol or streptomycin) by directly observed therapy (DOT).
   * The induction regimen:

     1. Induction regimens must have at least 40 DOT doses (if daily) or at least 56 DOT daily dose equivalents (if twice weekly). No more than 2 of every 7 total doses may be self-administered. Total induction doses (both DOT and self-administered) should not exceed 70. Induction should be completed within 12 weeks
     2. The ethambutol or streptomycin may be discontinued if the patient continues on adequate induction therapy with INH, rifampin and PZA, and if the M. tuberculosis isolate is susceptible to INH and rifampin.
   * If this induction regimen is not tolerated by the patient, a rifampin-containing regimen compatible with CDC/ATS recommendations is an acceptable alternative.
4. Age 18 years or older
5. Willingness to practice effective contraception (if female and of child-bearing potential)
6. Provision of written informed consent. Signed by both the patient and investigator, in accordance with Institutional Review Board requirements

Exclusion Criteria:

* Treatment with a drug(s) with high anti-mycobacterial activity for more than 15 days in the two months PRIOR to the start of anti-tuberculosis treatment, unless co-enrolled in TBTC Study 23, TBTC Study 24 or another TBTC treatment study.
* Patients with only extrapulmonary tuberculosis, unless co-enrolled in TBTC Studies 23, TBTC Study 24, or another TBTC treatment study.
* Skeletal tuberculosis
* Silicotuberculosis
* Patient intolerance of rifamycins, or MTB resistance to rifamycins
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pulmonary TB suspects
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Marc Weiner, MD, Principal Investigator — Audie L. Murphy VA Hospital
Locations (14):
- United States (10):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Chicago-Lakeside VAMC, Chicago, Illinois
  - Harlem Hospital Center, New York, New York
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
- Nelson R. Mandela School of Medicine, Durban, KwaZulu-Natal, South Africa
- Makerere University Medical School, Kampala, Uganda

REFERENCES:
- See also: (Click here for more information about the Tuberculosis Trials Consortium(TBTC) — http://www.cdc.gov/nchstp/tb/tbtc/